CLINICAL TRIAL: NCT02433197
Title: Effectiveness of an Individualized Program of Muscular Strength and Endurance Program With Aerobic Training for Improving Germ Cell Cancer Related Fatigue in Men Undergoing Chemotherapy
Brief Title: Effectiveness of an Individualized Program of Muscular Strength and Endurance Program for Improving Germ Cell Cancer
Acronym: EFICATEST
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Dr. Antonio I Cuesta-Vargas, Professor of Faculty of Health Sciences, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FCCSS-UMA_04-15
Record Dates: First submitted 2015-04-13; First posted 2015-05-04 (Estimated); Last update posted 2023-12-01 (Actual); Status verified 2017-03

CONDITIONS: Testicular Germ Cell Cancer
Keywords: Testicular cancer; Germ cell cancer; Physical exercise; Cancer-related fatigue; Chemotherapy; Clinical rules; Metabolomics
MeSH Terms: conditions — Testicular Neoplasms; Neoplasms, Germ Cell and Embryonal; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aerobic program (Experimental): Individualized physiotherapy strength and muscular endurance with aerobic training, led by physiotherapists in groups of 8-10 participants.
  Interventions: Device: Aerobic program
- Control group (No Intervention): They will be instructed to continue their current activities and not to increase objectively levels of physical activity performed during the 8-week intervention.

INTERVENTIONS:
Device: Aerobic program — The intervention will be an 8-week program of individualized physiotherapy strength and muscular endurance with aerobic training, led by physiotherapists in groups of 8-10 participants. Each program will be individualized based on the evaluations of muscular strength and enduranceas well as determination of aerobic-anaerobic zone transition described in previous studies In sessions of one hour 3 times a week. Each session will consist of 30 minutes of exercises performed on land followed by 20 minutes of continuous running in treadmill.
  In week 1 and 2 participants carry out 3 sets of 15 repetitions (reps) to become familiar with the exercises. From week 3 onwards participants will perform 4 sets of 10 reps. If the participant can do more than 12 reps, weight will be increased. All exercises are conducted supervised to ensure proper technique and adequate progression.
  Arms: Aerobic program

SUMMARY:
Background: Patients with testicular germ cell cancer (GCC) have a high cure rate, however impaired muscle function and fatigue are the most common complications among patients with GCC undergoing treatment with chemotherapy. Although exercise is widely recommended, information about physiopathological effects of cancer therapy in skeletal muscle is very limited.

Methods/Design: The present study is a randomized controlled trial comparing an individualized program of muscular strength and endurance with aerobic training compared to a control group. All variables will be measured at the beginning and at the end of a 8-week intervention by the same evaluator, who will hide the disposition of participants to each group. Besides, it will be monitoring during de following 6 months (24 weeks) after training for all outcome variables.

DETAILED DESCRIPTION:
Background: Patients with testicular germ cell cancer (GCC) have a high cure rate, however impaired muscle function and fatigue are the most common complications among patients with GCC undergoing treatment with chemotherapy. Although exercise is widely recommended, information about physiopathological effects of cancer therapy in skeletal muscle is very limited. Our aim is to evaluate the effects of an individualized exercise program with aerobic training in water running on cancer-related fatigue.

Methods/Design: The present study is a randomized controlled trial comparing an individualized program of muscular strength and endurance with aerobic training compared to a control group. The investigators will conduct this trial in patients undergoing chemotherapy, recruited by the Departament of Oncology of Virgen de la Victoria Hospital (Málaga). Patients will be included and evaluated before the first cycle of chemotherapy and assigned experimental or control group randomly. All variables will be measured at the beginning and at the end of a 8-week intervention by the same evaluator, who will hide the disposition of participants to each group. Besides, it will be monitoring during de following 6 months (24 weeks) after training for all outcome variables.

ELIGIBILITY:
Inclusion Criteria:

* Patients programmed to chemotherapy

Exclusion Criteria:

-

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-12 (Actual); Primary Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Cancer-related fatigue QuickPiper scale | 20 minutes
  The primary outcome will be fatigue, assessed by the revised Cancer-related fatigue QuickPiper scale, with the semi-structured interview used by Cella et al (1998) to define phenotype of CRF

SECONDARY OUTCOMES:
Sf-12 | 10 min
  The state of physical and mental health
EuroQoL-5D | 10 min
  Quality of life
Profile of Mood States | 10 min
  It is possible to obtain an overall index of altered mood and seven partial measures: stress / anxiety, depression / rejection, anger / hostility, vigor / activity, fatigue / inertia and confusion / bewilderment
Physical condition test | 20 min
  strength peak of knee extension (quadriceps), knee flexion (hamstring), elbow extension (brachial triceps) and elbow flexion (biceps brachii) by one dynamometry instrumented with Powertruck II of JTECH, following the protocol described by Daniels & Worthingham (1995). Hand grip strength will be evaluated by the hydraulic dynamometer JAMAR
C-reactive protein (CRP) | 20 min
  It will be measured in blood samples following clinical standards in 10 ml venous blood
Tumor Necrosis Factor alpha (TNF-a) | 20 min
  It will be measured in blood samples following clinical standards in 10 ml venous blood sample.
Interleukin-6 (IL-6), Interleukin-18 (IL-18), Interleukin-4 (IL-4) and Interleukin-10 (IL 10) | 20 min
  It will be measured in blood samples following clinical standards in 10 ml venous blood
high density lipoprotein (HDL), low density lipoprotein (LDL) cholesterol, triglycerides | 20 min
  It will be measured in blood samples following clinical standards in 10 ml venous blood

CONTACTS AND LOCATIONS:
Overall Officials: Antonio I Cuesta-Vargas, Study Director — University of Malaga
Locations (1):
- Antonio Cuesta-Vargas, Málaga, Spain

REFERENCES:
- [Derived] Cuesta-Vargas AI, Carabantes F, Caracuel Z, Conejo I, Alba E. Effectiveness of an individualized program of muscular strength and endurance with aerobic training for improving germ cell cancer-related fatigue in men undergoing chemotherapy: EFICATEST study protocol for a randomized controlled trial. Trials. 2016 Jan 5;17:8. doi: 10.1186/s13063-015-1143-x. PMID 26732120